CLINICAL TRIAL: NCT02970851
Title: Effect of Endothelin Receptor Antagonist Bosentan in Glucose Metabolism of the Myocardium and Coronary Dependant Endothelial Vasoreactivity Measured by 18F-FDG PET / CT and 82Rb PET / CT in Patients With PAH or CTEPH
Brief Title: Bosentan in Myocardium Metabolism and Perfusion Measured by 18F-FDG and 82Rb PET/CT on PAH and CTEPH
Status: Terminated | Type: Observational
Why Stopped: Slow patient recruitment after arrival of macitentan on the market
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, John O. Prior, Chief of the Department of Nuclear medicine, University of Lausanne Hospitals
Other Study IDs: 08/12
Record Dates: First submitted 2016-06-19; First posted 2016-11-22 (Estimated); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Myocardial Dysfunction; Endothelial Dysfunction
Keywords: Endothelin receptor antagonist (ERA); pulmonary artery hypertension (PAH),; 18F-2-fluoro-2-deoxy-D-glucose (18F-FDG) PET/CT; Rubidium-82 (82Rb) PET/CT
MeSH Terms: conditions — Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess the effect of bosentan on the myocardial metabolism and the dependent endothelial coronary vasomotoricity in patients presenting a PAH.

Hypothesis : Bosentan may improve right ventricular function by decreasing myocardial stress and glucose metabolism. Patients may benefit from images with 18F-FDG PET / CT and 82Rb PET / CT for an earlier assessment and optimal management of PAH.

DETAILED DESCRIPTION:
Patients refered to the hospital for a right heart catheterization for a PAH suspected at the echocardiography will be presented with the protocol.If inclusion/exclusion criteria are fulfilled all the procedures will be planned. At the screening visit the patient will have a right heart catheterization and an echocardiography. After a maximum of 4 weeks each patient will have 18F-FDG and 82Rb PET/CTs before start of treatment with Bosentan. These PET/CTs together with an echocardiography will be repeated at 6 and 12 weeks after start of treatment with bosentan.

Finally a right heart catheterization will be planned at 12 weeks after start of treatment with bosentan as a routine procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic PAH (PH group 1 Dana Point / stages 2 à 4 according to NYHA classification, defined by a mean arterial pulmonary pressure >25 millimeter of mercury (mmHg) at rest, an occlusion arterial pulmonary pressure <15 millimeter of mercury (mmHg) and vascular pulmonary resistance >240 dyn.s.cm-5 for which a treatment with bosentan is indicated Or Patients with CTEPH not candidate for a pulmonary endarterectomy or patient with residual CTEPH after pulmonary endarterectomy (PH group 4 Dana Point / stages 2 to 4 according to NYHA classification) and for which a treatment with bosentan is indicated
* Indication to perform a right heart catheterization in the context of PAH suspected during cardiac ultrasound
* Age from 18 to 80 years old, male and female
* Karnofsky index ≥80%
* Informed consent signed

Exclusion Criteria:

* Patients with PAH stages 2,3 or 5 of Dana Point
* Patients with a contra-indication to adenosine including severe uncontrolled asthma, severe uncontrolled chronic obstructive pulmonary disease, 2nd or 3rd degree atrioventricular block without pacemaker,
* Patients with a contraindication to Bosentan, i.e :hypersensibility to the product, hepatic failure Child Pugh B or C, aminotransferases >3 times normal value (N),association with cyclosporine A or glibenclamide
* Pregnancy, female of child-bearing potential not using any acceptable contraceptive method, breastfeeding
* Atrial fibrillation (Ventricular Ejection Fraction (VEF) not evaluable at echography)
* Karnofsky index <80%
* Impossibility to obtain informed consent signed
* Left cardiopathies that can be responsible of post-capillar hypertension
* Involvement in another clinical study with an unregistered drug within 30 days prior to this specific study and during the entire course of the study
* Inability to comply with study procedures (linguistic problem, psychiatric problems, dementia, confusional state)
* Known or suspected non compliance drug or alcohol abuse
* Left heart assessment : diastolic and systolic function and valvular structures to exclude a cardiac pathology

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients eligible for Bosentan therapy
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Analysis of each method of imaging for assessment of myocardial metabolism | Baseline
  On the images of au 18F-FDG PET/CT : myocardial ventricular right maximum standardized uptake value (SUVmax)
Analysis of each method of imaging for assessment of myocardial metabolism | at 4 weeks after start of treatment
  myocardial ventricular right maximum standardized uptake value (SUVmax) on the images of au 18F-FDG PET/CT
Analysis of each method of imaging for assessment of myocardial metabolism | at 6 weeks after start of treatment
  On the images of au 18F-FDG PET/CT : myocardial ventricular right maximum standardized uptake value (SUVmax)
Analysis of each method of imaging for assessment of myocardial metabolism | at 12 weeks after start of treatment
  On the images of au 18F-FDG PET/CT : myocardial ventricular right maximum standardized uptake value (SUVmax)
On the images 82Rb PET/CT rest MBF | Baseline
  myocardial blood flow (MBF in mL/min/g) at rest
On the images 82Rb PET/CT rest MBF | at 4 weeks after start of treatment
  myocardial blood flow (MBF in mL/min/g) at rest
On the images 82Rb PET/CT rest MBF | at 6 weeks after start of treatment
  myocardial blood flow (MBF in mL/min/g) at rest
On the images 82Rb PET/CT rest MBF | at 12 weeks after start of treatment
  myocardial blood flow (MBF in mL/min/g) at rest
On the images 82Rb PET/CT stress MBF | Baseline
  myocardial blood flow (MBF in mL/min/g) at pharmacological stress
On the images 82Rb PET/CT stress MBF | at 4 weeks after start of treatment
  myocardial blood flow (MBF in mL/min/g) at pharmacological stress
On the images 82Rb PET/CT stress MBF | at 6 weeks after start of treatment
  myocardial blood flow (MBF in mL/min/g) at pharmacological stress
On the images 82Rb PET/CT stress MBF | at 12 weeks after start of treatment
  myocardial blood flow (MBF in mL/min/g) at pharmacological stress
On the images 82Rb PET/CT, analysis of endothelial dysfunction cold test MBF | Baseline
  myocardial blood flow (MBF in mL/min/g) at cold test
On the images 82Rb PET/CT, analysis of endothelial dysfunction cold test MBF | at 4 weeks after start of treatment
  myocardial blood flow (MBF in mL/min/g) at cold test
On the images 82Rb PET/CT, analysis of endothelial dysfunction cold test MBF | at 6 weeks after start of treatment
  myocardial blood flow (MBF in mL/min/g) at cold test
On the images 82Rb PET/CT, analysis of endothelial dysfunction cold test MBF | at 12 weeks after start of treatment
  myocardial blood flow (MBF in mL/min/g) at cold test
Analysis of each method of imaging for assessment of myocardial metabolism and endothelial dysfunction | Baseline
  On the images of au 18F-FDG PET/CT : myocardial ventricular left maximum standardized uptake value (SUVmax)
Analysis of each method of imaging for assessment of myocardial metabolism and endothelial dysfunction | at 4 weeks after start of treatment
  On the images of au 18F-FDG PET/CT : myocardial ventricular left maximum standardized uptake value (SUVmax)
Analysis of each method of imaging for assessment of myocardial metabolism and endothelial dysfunction | at 6 weeks after start of treatment
  On the images of au 18F-FDG PET/CT : myocardial ventricular left maximum standardized uptake value (SUVmax)
Analysis of each method of imaging for assessment of myocardial metabolism and endothelial dysfunction | at 12 weeks after start of treatment
  On the images of au 18F-FDG PET/CT : myocardial ventricular left maximum standardized uptake value (SUVmax)

SECONDARY OUTCOMES:
Analysis of right heart catheterization parameters PAP | at screening
  pulmonary arterial pressure (PAP)
Analysis of right heart catheterization parameters PAP | at 12 weeks after start of treatment
  PAP
Analysis of right heart catheterization parameters RAP | at screening
  right atrial pressure (RAP)
Analysis of right heart catheterization parameters RAP | at 12 weeks after start of treatment
  RAP
Analysis of right heart catheterization parameters PWP | at screening
  pulmonary wedge pressure (PWP)
Analysis of right heart catheterization parameters PWP | at 12 weeks after start of treatment
  PWP
Analysis of clinical parameters NYHA | at screening
  NYHA classification
Analysis of clinical parameters NYHA | at 12 weeks after start of treatment
  New York Heart Association (NYHA) classification
Analysis of clinical parameters 6-min walk test | at screening
  6-minute walk test
Analysis of clinical parameters 6-min walk test | at 12 weeks after start of treatment
  6-minute walk test
Analysis of clinical parameters LFT | at screening
  Results of lung function tests
Analysis of clinical parameters LFT | at 12 weeks after start of treatment
  Results of lung function tests
Analysis of clinical parameters NT-pro-BNP | at screening
  plasmatic N terminal - pro - Brain Natriuretic Peptide (NT-pro-BNP)
Analysis of clinical parameters NT-pro-BNP | at 12 weeks after start of treatment
  plasmatic NT-pro-BNP

CONTACTS AND LOCATIONS:
Overall Officials: John O Prior, MD PhD, Principal Investigator — Lausanne University Hospitals
Locations (1):
- Centre Hospitalier Universitaire Vaudois, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: abstract poster presentation about present study — https://erj.ersjournals.com/content/50/suppl_61/PA2414